CLINICAL TRIAL: NCT07171723
Title: Effects of Antagonizing the Ghrelin Receptor in Individuals With Obesity on Treatment With Semaglutide
Brief Title: Studying the Influence of LEAP2 on Integrated Endocrine Control of Eating During Semaglutide Treatment
Acronym: SILENCED
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Asger Lund, MD, MD, Ph.d, Head of Department, Center for Clinical Metabolic Research, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-25035700
Record Dates: First submitted 2025-09-08; First posted 2025-09-12 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Obesity &Amp; Overweight
MeSH Terms: conditions — Obesity; Overweight | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LEAP2 (Experimental): An intravenous infusion of LEAP2, an endogenous inverse agonist and competitive antagonist of the ghrelin receptor (GHSR), will be administered at 40 pmol/kg/min for 6 hours.
  Interventions: Biological: Liver-Expressed Antimicrobial Peptide 2 (LEAP2)
- Placebo (Placebo Comparator): An intravenous infusion of isotonic saline (placebo) will be administered for 6 hours
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Biological: Liver-Expressed Antimicrobial Peptide 2 (LEAP2) — Continuous intravenous infusion of LEAP2 (Liver-Expressed Antimicrobial Peptide 2), an endogenous inverse agonist and competitive antagonist of the ghrelin receptor (GHSR), administered at 40 pmol/kg/min for 6 hours. LEAP2 inhibits ghrelin-mediated signaling involved in hunger regulation, gastric motility, and growth hormone secretion. This intervention enables investigation of the physiological relevance of ghrelin receptor activity during semaglutide-induced appetite suppression
  Arms: LEAP2
Other: Placebo (saline) — Continuous intravenous infusion of isotonic saline (0.9% sodium chloride) for 6 hours. This placebo comparator is used to match the volume, rate, and duration of the active intervention (LEAP2) in a randomized, double-blind, crossover design. The placebo enables assessment of the physiological effects of ghrelin receptor blockade by LEAP2 in individuals with obesity treated with semaglutide
  Arms: Placebo

SUMMARY:
This clinical study investigates how blocking the hunger-related ghrelin receptor affects appetite and metabolism in individuals with obesity who are treated with semaglutide (a GLP-1 receptor agonist). LEAP2, a naturally occurring hormone that inhibits the ghrelin receptor, is used as the investigational compound. The objective of the study is to clarify how the ghrelin system functions when appetite is suppressed by semaglutide treatment. Participants will receive either LEAP2 or placebo during two experimental visits in a randomized, double-blind, crossover design. The investigators will assess food intake, appetite sensations, glucose metabolism, and hormonal responses. By examining the interaction between semaglutide and ghrelin signaling, the study aims to improve understanding of how multiple appetite-regulating systems interact and whether additional hunger signals remain active during GLP-1 treatment. The findings may inform the development of future treatments for individuals with obesity.

DETAILED DESCRIPTION:
This study investigates the physiological role of ghrelin receptor signaling in individuals with obesity receiving stable treatment with semaglutide, a glucagon-like peptide-1 (GLP-1) receptor agonist known to suppress appetite and induce weight loss. Ghrelin is the only known circulating orexigenic gut hormone, and its activity is mediated via the growth hormone secretagogue receptor (GHSR). Whether ghrelin signaling continues to contribute meaningfully to appetite regulation during pharmacological GLP-1 receptor activation remains unknown.

Liver-expressed antimicrobial peptide 2 (LEAP2) is an endogenous inverse agonist and competitive antagonist of the GHSR. LEAP2 provides a highly specific and transient means of blocking ghrelin receptor activity in humans, enabling mechanistic exploration of its physiological relevance. Previous studies have demonstrated that LEAP2 infusion reduces ad libitum food intake and postprandial glucose excursions in both lean and obese individuals. However, the role of ghrelin signaling under conditions of GLP-1-induced appetite suppression has not been elucidated.

The SILENCED study is a randomized, double-blind, placebo-controlled, crossover trial. Twenty-four participants with obesity who are weight-stable and on a stable dose of ≥1 mg/week semaglutide for at least 3 months will complete two experimental study days. Each participant will receive a 6-hour intravenous infusion of either LEAP2 or placebo (saline) on separate days. During each visit, appetite-related measures, food intake, glucose metabolism, gastrointestinal motility, growth hormone levels, and energy expenditure will be assessed.

The primary outcome is total energy intake during a standardized ad libitum meal. Secondary and exploratory outcomes include visual analogue scale ratings of appetite, gastric emptying assessed via paracetamol absorption, postprandial glucose and hormone responses, and indirect calorimetry measurements.

This study is expected to provide novel insight into whether ghrelin receptor signaling continues to play a functional role in appetite and metabolism under pharmacological GLP-1 receptor activation. The findings may inform the development of future combination therapies targeting multiple appetite-regulating pathways in the treatment of obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Body mass index (BMI) above ≥ 25 kg/m2
* Ongoing semaglutide treatment with a stable dose of ≥ 1 mg once weekly for a minimum of 3 months prior to inclusion
* Weight stability, defined as a maximum variation of ±3% between the highest and lowest recorded body weight during the 3 months prior to inclusion.
* Informed oral and written consent

Exclusion Criteria:

* Anaemia
* Alanine aminotransferase (ALAT) > 2 times normal value
* History of hepatobiliary and/or gastrointestinal disorder
* Kidney disease (serum creatinine above normal range and/or urine albumin-creatinine ratio 30mg/g confirmed with two measurements)
* Any ongoing medication that investigator evaluates would interfere with study participation
* Any physical or psychological condition that investigators evaluate would interfere with study participation including any acute or chronic illnesses.
* Regular tobacco smoking and/or use of other nicotine products
* Glycated haemoglobin HbA1c > 48 and/or type 1 or type 2 diabetes medical treatment
* Women of childbearing potential who are not using effective contraception
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Food intake | 290 to 310 minutes
  Difference in total energy intake during a standardized ad libitum meal. Energy intake will be quantified as kilojoules (kJ) and kJ per kilogram of body weight consumed during the meal

SECONDARY OUTCOMES:
Composite score of sensation of hunger, fullness (reverse corded) and prospective food intake. | -30 to 290 minutes
  Visual analogue scales (VASs) assessing appetite, satiety and hunger sensations (from 0 to 10 cm on a scale = from mimimum to maximum sensation)
Gastric emptying | -30 to 290 minutes
  Paracetamol concentration in plasma after intake of 1.5 g paracetamol
Plasma concentrations of glucose | -30 to 290 minutes
  Plasma glucose
Circulating levels of growth hormone and IGF-1 | -30 to 290 minutes
  Blood samples
Circulating levels of acyl-ghrelin | -30 to 290 minutes
  Blood samples

OTHER OUTCOMES:
Sensation of nausea, thirst, and comfort | -30 to 290 minutes
  VAS
Circulating levels of LEAP2, insulin, glucagon, and other hormones and signaling molecules regulating glucose metabolism, gastrointestinal motility, energy expenditure and eating behaviour | -30 to 290 minutes
  Blood samples
Lipids and other metabolism markers | -30 to 290 minutes
  Blood samples
Energy expenditure | -30 to 290 minutes
  Indirect calorimetry
Duration of ad libitum meal | 290 to 310 minutes
  Ad libitum meal duration
Water intake during ad libitum meal | 290 minutes to 310 minutes
  Ad libitum meal
Water intake during ad libitum meal | 290 to 310 minutes
  Ad libitum meal water-intake
Gallbladder motility | 290 to 310 minutes
  Bed-side ultrasonography
Systolic and diastolic blood pressure | -30 to 290 minutes
  Blood pressure measurement
Heart rate | -30 to 290 minutes
  Heart rate measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
At this stage, no final decision has been made regarding sharing of individual participant data (IPD). While sharing de-identified data could contribute to scientific transparency, reproducibility, and collaborative advancement in obesity and metabolic research, several factors must be considered. These include ethical and legal obligations related to participant confidentiality, the need for appropriate data-use agreements, and institutional policies on data governance. The possibility of sharing IPD will be revisited upon study completion, in alignment with sponsor requirements, ethical approvals, and journal publication policies